CLINICAL TRIAL: NCT01095640
Title: A Multicenter, Double-Blind, Randomized, Vehicle-Controlled, Parallel Group Study Comparing 0.3% Adapalene Topical Gel (Actavis Mid Atlantic LLC) to Differin® (0.3 % Adapalene Topical Gel) (Galderma Laboratories, L.P.) and Both Active Treatments to a Vehicle Control (Actavis Mid Atlantic LLC) in the Treatment of Mild to Moderate Acne Vulgaris
Brief Title: Study Comparing 0.3% Adapalene Topical Gel to Differin® 0.3% Adapalene Topical Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actavis Mid-Atlantic LLC (Industry)
Responsible Party: Christine M. Winslow, Ph.D., Director Clinical Development, Actavis Mid-Atlantic LLC
Organization: Actavis Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADAP-0.3/2008
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Acne Vulgaris
Keywords: acne; adapalene; Differin
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- adapalene 0.3% topical gel (Actavis Mid-Atlaqntic LLC) (Experimental)
  Interventions: Drug: adapalene 0.3% topical gel
- Differin® (adapalene 0.3% topical gel) (Active Comparator)
  Interventions: Drug: adapalene 0.3% topical gel
- Vehicle Control (Placebo Comparator)
  Interventions: Drug: adapalene 0.3% topical gel

INTERVENTIONS:
Drug: adapalene 0.3% topical gel — once a day, 84 days

SUMMARY:
Marketed by Galderma Laboratories, L.P., Differin® (adapalene 0.3% topical gel) is a safe and effective topical therapy used for the treatment of acne vulgaris. Actavis Mid-Atlantic LLC has developed a generic formulation of adapalene 0.3% topical gel and the current study is designed to evaluate the safety and efficacy of this formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients must be 12 years old or older.
2. Patients who are 18 years of age or older must have provided IRB approved written informed consent. Patients between the ages of 12 to 17 years of age must have provided IRB approved written assent; this written assent must be accompanied by an IRB approved written informed consent from the patient's legally acceptable representative (i.e., parent or guardian). In addition, all patients or their legally acceptable representatives (i.e., parent or guardian) must sign a HIPAA authorization, if applicable
3. Patients must have a definite clinical diagnosis of acne vulgaris of mild to moderate severity (Grade 2 or Grade 3 on the IGE).
4. Patients must have a minimum of 20 and a maximum of 60 facial inflammatory lesions at baseline. Patients must also have a minimum of 20 and a maximum of 75 facial comedones at baseline. Patients may have no more than one (1) nodulo-cystic lesion at baseline. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area. Lesions involving the eyes, angles of the nose (i.e., the lines around your nostrils and under the nostrils) and scalp should be excluded from the count. Patients may have acne lesions on other areas of the body (e.g., on the back).
5. Female patients of childbearing potential must have been using and must agree to continue to practice abstinence or use accepted methods of birth control, from 30 days prior to study entry to 30 days after the last administration of study drug. All female patients are considered to be of childbearing potential unless they have been surgically sterilized or have been postmenopausal for at least 1 year. Abstinence is an acceptable method of birth control. Alternatively, any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®) Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD. Female patients must have a negative urine pregnancy test at baseline.
6. All male patients must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Alternatively, any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®), Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD.
7. Patients must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.
8. Patients must be willing to refrain from using any treatments for acne vulgaris, other than the investigational product, for acne present on the face. Patients may use other topical acne treatments that do not have significant or measurable systemic absorption for treatment of acne of the back, shoulders and chest (e.g., benzoyl peroxide, salicylic acid).
9. Patients must be in good health and free from any clinically significant disease, including but not limited to, conditions that may interfere with the evaluation of acne vulgaris. Such conditions include, but are not limited to the following: rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne; carcinoid syndrome; mastocytosis; acneiform eruptions caused by make-up, medication, facial psoriasis and facial eczema.
10. Patients who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.

Exclusion Criteria:

1. Female patients who are pregnant, nursing or planning to become pregnant during study participation (Visit 1 through Visit 5 or Early Discontinuation Visit) will be excluded from study participation.
2. Patients who have a known hypersensitivity to adapalene and its excipients will be excluded from study participation.
3. Patients who have acne congoblata, acne fulimans, and secondary acne (e.g., chloracne and drug induced acne) will be excluded from participation.
4. Patients who have been treated with systemic antibiotics or systemic anti-acne drugs within 30 days prior to baseline will be excluded from study participation.
5. Patients who have been treated with prescription and/or over-the-counter topical medications for the treatment of acne vulgaris including antibiotics, topical corticosteroids or topical anti-inflammatory medications on the face within 14 days prior to baseline will be excluded from study participation.
6. Patients who are currently taking or have been treated with corticosteroids (including intranasal or inhaled corticosteroids) within 30 days prior to baseline will be excluded from study participation.
7. Patients who have started hormonal therapy or changed the dosage of their hormonal therapy within 30 days prior to baseline will be excluded from study participation. The dosage and frequency of use of any hormonal therapy started greater than 30 days prior to baseline must remain unchanged throughout the study (Visit 1 through Visit 5 or Early Discontinuation Visit). Hormonal treatments include, but are not limited to, estrogenic and progestational agents such as birth control pills.
8. Patients who have received oral retinoids (e.g., isotretinoin) within 180 days prior to study entry or have applied topical retinoids (e.g., tretinoin, tazarotene, adapalene) to the face within the 30 days prior to baseline will be excluded from study participation.
9. Patients who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline will be excluded from study participation.
10. Patients who have unstable medical disorders that are clinically significant or life-threatening diseases will be excluded from study participation.
11. Patients who have on-going malignancies requiring systemic treatment will be excluded from study participation. In addition, patients who have any malignancy of the skin of the facial area will be excluded from study participation.
12. Patients who have facial hair will be excluded from study participation. Unacceptable facial hair includes, but is not limited to, beards and long side-burns. A well-trimmed mustache is acceptable. Patients who have performed wax epilation of the face within 14 days prior to baseline will also be excluded from study participation.
13. Patients who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold, will be excluded from study participation.
14. Patients who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids, cocaine and barbiturates)as judged by history will be excluded from study participation.
15. Patients who have participated in an investigational drug study (i.e., patients have been treated with an investigational drug) within 30 days prior to baseline will be excluded from study participation. Patients who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
16. Patients who have been previously enrolled in this study will be excluded from study participation.
17. Patients who have had laser therapy, electrodessication and phototherapy (e.g., ClearLight®) to the facial area within 180 days prior to study entry will be excluded from participation.
18. Patients who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry will be excluded from participation.
19. Patients who currently have or have recently had bacterial folliculitis will be excluded from participation.
20. Patients who have a baseline local irritation score of 3 (severe, marked/intense) as scored using the Local Irritation Scale (Section 5.2) will be excluded from participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1159 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Therapeutic Equivalence | 12 weeks
  The primary equivalence comparison is that between the test and reference products for the mean percent change from baseline in the inflammatory lesion counts, the non-inflammatory lesion counts and the proportion of "success" patients at Visit 5, as measured using the Investigator's Global Evaluation (IGE).
Superiority | 12 Weeks
  The primary superiority evaluations are the comparisons between each active treatment and the vehicle control relative to the mean percent change in the inflammatory lesion counts, the non-inflammatory lesion counts and the proportion of "success" patients at Visit 5, as measured using the IGE.
Safety | 12 Weeks
  All treatment-emergent adverse events reported during the study will be summarized in order to assess safety.

SECONDARY OUTCOMES:
Total Lesions | 12 Weeks
  The secondary efficacy measure is the mean percent reduction in the total lesion count (inflammatory lesion count + non-inflammatory lesion count) at Visit 5.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal B., MD, Principal Investigator — Yenepoya Medical College; Bela J. Shah, MD, Principal Investigator — GMC and SSG Hospital; Mhaske, MD, Principal Investigator — B. J. Medical College and Hospital; Manoj K. Parekh, MD, Principal Investigator — Bhagwan Mahaveer Jain Hospital; V. R. Sardesai, MD, Principal Investigator — Bharati Vidyapeeth University Medical College & Hospital; Kailash Bhatia, MD, Principal Investigator — Bhatia Skin Laser & Cosmetic Centre; Leelavathy B., MD, Principal Investigator — Bowring & Lady Curzon Hospital; Rajkumar V., MD, Principal Investigator — Dhanawantari Polyclinic; Mukta Sachdev, MD, Principal Investigator — Dr. Mukta Skin Clinic; Anilkumar Malik, MD, Principal Investigator — G.M Modi Hospital; Yogesh Marfatia, MD, Principal Investigator — GMC and SSG Hospital; Mahendra M. Kura, MD, Principal Investigator — Grant Medical College & Sir JJ Group of Hospitals; Jayadev Betkerur, MD, Principal Investigator — J.S.S. Medical College Hospital; Manjunath S. M., MD, Principal Investigator — Justice K.S. Hegde Charitable Hospital; Ramesh M., MD, Principal Investigator — Kempegowda Institute of Medical Sciences; Hemanji R. Jerajani, MD, Principal Investigator — L.T.M. Medical College & General Hospital; Vijaykumar Garg, MD, Principal Investigator — Maulana Azad Medical College Hospital; Rajitha K., MD, Principal Investigator — Medwin Hospital; Putta Srinivas, MD, Principal Investigator — Osmania General Hospital; Alur S. Kumar, MD, Principal Investigator — Owaisi Hospital & Research Centre; Jayesh Kothari, MD, Principal Investigator — Skin Clinic; P. V. S. Prasad, MD, Principal Investigator — Rajah Muthiah Medical College Hospital; D. N. Balraj, PI, Principal Investigator — Rajbal Skin Clinic; Sailaja K. Surapaneni, MD, Principal Investigator — SRI Medical Aesthetic and Cosmetic Surgery; Ravi M. Rathod, MD, Principal Investigator — Skin Care Centre; Ranjan C. Raval, MD, Principal Investigator — Smt. NHL Medical College and V.S. Hospital; V. K. Somani, MD, Principal Investigator — Somani Skin and Cosmetology Institute; Rachita Dhurat, MD, Principal Investigator — T. N. Medical College and BYL Nair hospital; P. V. Patalay, MD, Principal Investigator — Vani Skin Clinic; Nataraja, MD, Principal Investigator — Victoria Hospital; Karigi Siddalingappa, MD, Principal Investigator — Vijayanagara Institute Of Medical Sciences
Locations (1):
- L.T.M. Medical College & General Hospital, Mumbai, India